CLINICAL TRIAL: NCT06423560
Title: Evaluation of Pulmonary Fibrosis After Severe Interstitial Pneumonia Due to COVID-19 (SARS-CoV-2)
Brief Title: Pulmonary Fibrosis After Severe COVID-19 Pneumonia
Acronym: SPIFFERO
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gabriele Fragasso, Principal Investigator, IRCCS San Raffaele
Other Study IDs: CET 145-2024
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Fibrosis; COVID-19
Keywords: COVID-19; Pulmonary fibrosis; ARDS; Computed tomography; pulmonary function test
MeSH Terms: conditions — Pulmonary Fibrosis; COVID-19 | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residual disease > 20% of the total lung volume was considered pathological at follow-up CT
  Interventions: Radiation: Computed tomography
- Residual disease < 20% of the total lung volume was considered pathological at follow-up CT
  Interventions: Radiation: Computed tomography

INTERVENTIONS:
Radiation: Computed tomography — Follow-up computed tomography at 3-6 months and 12 months
  Other Names: Pulmonary function test; Echocardiography

SUMMARY:
Patients discharged after hospitalization for COVID-19 pneumonia were retrospectively selected by radiologically established criteria that at admission presented at chest computed tomography (CT) (i) normal lung parenchyma <50% of total lung volume; and/or (ii) area of lung consolidation > 10%. All At discharge and after 9 months, all subjects underwent cardiological evaluation, echocardiogram, pulmonary function tests (PFT) both atby 3 and by 12 months after discharge. Chest CT was performed by 12 months after discharge and chest CT. Specifically, the magnitude of pulmonary involvement between baseline and follow-up was considered the primary endpoint of this study. Secondary endpoints of the study were results of respiratory function testing, echocardiographic parametersparameters, and persistence of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Hospitalization for severe COVID-19 pneumonia
* Computed tomography during index hospitalization that showed: (i) normale lung parenchyma < 50% of total lung volume and/or (ii) parenchymal consolidation > 10%
* Cardiological and pneumological visit, echocardiography and pulmonary function test at 3 and 12 months from hospital discharge
* Computed tomography by 12 months from hospital discharge

Exclusion Criteria:

* Age < 18
* Absence of previously cited test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for sever COVID-19 pneumonia and successively discharge and with a 1-year follow-up
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
The magnitude of pulmonary involvement | 12 months

SECONDARY OUTCOMES:
results of respiratory function testing | 12 months
echocardiographic parameters | 12 months
persistence of symptoms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fragasso, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided